CLINICAL TRIAL: NCT07148479
Title: Comparison of Telerehabilitation and Traditional Balance Training in Post Menopausal Women With Osteoporosis.
Brief Title: Telerehabilitation Versus Traditional Balance Training in Women With Osteoporosis.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Mehak bibi
Record Dates: First submitted 2025-08-24; First posted 2025-08-29 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Osteoporosis Postmenopausal
Keywords: Telerehabilitation; Balance; Osteoporosis; Posmenopausal; Virtual exercise
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis

STUDY DESIGN:
Intervention Model Description: There will be comparison between the two groups, experimental and control.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation group (Experimental): This group will receive a 6 week structured telerehabilitation exercise protocol of low to moderate intensity (18 sessions , 3 sessions per week,45 to 60 minutes ), warmup, balance training and cool down exercises. delivered online by a physiotherapist and progressively increasing every three weeks.
  Interventions: Other: Telerehabilitation group
- Traditional Balance Training group (Active Comparator): In the traditional balance training group the protocol will be delivered by a physiotherapist in a clinical environment face to face. The standardized balance training protocol will be monitored exactly the same as telerehabilitation group
  Interventions: Other: Traditional balance training group

INTERVENTIONS:
Other: Telerehabilitation group — The telerehabilitation group participated in balance training sessions delivered through secure virtual platforms such as WhatsApp video calls. Participants completed 3 sessions per week, each lasting 45-60 minutes, over a total of 6 weeks (18 sessions). The program target static, dynamic, anticipatory, and reactive balance. participants will use households items.session began with warm-up exercises such as gentle marching, arm circles, and hamstring stretches, followed by balance training targeting static, dynamic, anticipatory, and reactive components. Exercises included heel-to-toe standing, single-leg stance, tandem stance, obstacle walking, heel-to-toe walking, side stepping, functional reach, weight shifting, caregiver-assisted perturbations, and foam surface standing. All exercises were performed in 3 sets with specified holds or repetitions. Sessions concluded with cool-down activities including tricep stretches, forward bends, and deep breathing.
  Arms: Telerehabilitation group
Other: Traditional balance training group — Same as telerehabilitation group but it will concluded in a clinical setting.
  Arms: Traditional Balance Training group

SUMMARY:
Osteoporosis is a silent disease that leads to fractures, postural deformities, and impaired balance, especially in postmenopausal women. In Pakistan, prevalence is high, with 39% of women reported as severely osteoporotic. Postmenopausal women with osteoporosis and balance issues face increased fall risk due to poor bone density, weakened muscles especially in the lower limb band altered posture .Balance and strength training reduce fall risk, but access to in-person rehabilitation is limited. Telerehabilitation provides remote delivery of structured exercise programs and has shown positive outcomes in balance and bone health. Few studies, however, have compared telerehabilitation with conventional training across all balance domains. The goal of this randomized controlled trial is to compare the effect of Telerehabilitation and Traditional Balance Training in Post Menopausal Women with osteoporosis. Participants will be randomly assigned to one of the two groups, and both will receive an identical standardized balance training program . The results of this clinical trial will help evaluate how telerehabilitation can improve the balance of postmenopausal women with osteoporosis and improve health outcomes.

DETAILED DESCRIPTION:
Osteoporosis often remains undetected until fractures occur, typically involving the hip, wrist, or spine, and may also cause back pain, height loss, and kyphosis. Postmenopausal women face increased fall risk due to reduced bone density, weakened lower limb muscles, and altered posture. Many also develop fear of falling, which restricts activity and accelerates muscle weakness.

Globally, osteoporosis affects about 23.1% of women and 11.7% of men, with fragility fractures being a major cause of disability. In Pakistan, hospital-based findings show a high proportion of postmenopausal women as severely osteoporotic, with a strong link to fall-related injuries.

Exercise interventions, including balance, resistance, and weight-bearing training, are known to improve bone strength, postural control, and confidence by stimulating bone remodelling and enhancing musculoskeletal performance. Telerehabilitation, delivered via video conferencing, provides remote access to such programs and has demonstrated improvements in stability, weight-shifting, and functional balance.

However, most studies assess limited outcomes using tools like TUG or BBS, without addressing static, dynamic, anticipatory, and reactive balance together. Evidence largely comes from high-income countries, while data from resource-limited settings like Pakistan remain scarce. This trial seeks to evaluate telerehabilitation compared to traditional training across comprehensive balance domains in postmenopausal women with osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

* • Women diagnosed with osteopenia and osteoporosis at hip and lumbar spine through DEXA

  * Age 50-70 years
  * Have mobile phones and can communicate in video call
  * Have Balance score (21-44) on berg balance scale
  * A caregiver must be available to assist the participant during Tele sessions.

Exclusion Criteria:

* • Women with severe mobility impairments.

  * Women with cognitive conditions affecting participation.
  * Women with lower limb joint injury or surgery

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in Berg Balance Scale score | Baseline and 6 weeks
  The Berg Balance Scale (BBS) is a widely used clinical tool to assess static and dynamic balance in individuals, particularly older adults. It's a 14-item test that evaluates a person's ability to perform various balance-related tasks, such as sitting, standing, reaching, and turning. Each item is scored on a 0-4 scale, with 0 indicating the lowest level of function and 4 indicating the highest. The total score ranges from 0 to 56, with lower scores suggesting a higher risk of falls

SECONDARY OUTCOMES:
Change in Time up and Go test score | Baseline and 6 weeks
  The Timed Up and Go Test (TUG) is a simple yet widely validated tool used to assess mobility and fall risk. It measures how quickly an individual can rise from a chair, walk three meters, turn, walk back, and sit down
Functional reach test | Baseline and 6 weeks
  The Functional Reach Test (FRT) assesses how far an individual can reach forward while standing, without stepping or losing balance. It's particularly effective for identifying balance limitations in frail or elderly populations
Change in Push and release test score | Baseline and 6 weeks
  Push and Release Test is designed to measure reactive postural control by observing how a person recovers after being released from a supported backward lean.
Change in Single leg stance test score | Baseline and 6 weeks
  The Single Leg Stance Test (SLS) is a simple but powerful tool to evaluate balance and stability, particularly in older adults or individuals with conditions like osteoporosis. In this test, the person is asked to stand on one leg usually with eyes open and hands on hips while the clinician times how long they can maintain that position without support. It's an effective way to spot balance problems that could lead to falls

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Huma Riaz, Principal Investigator — Riphah International University
Locations (1):
- Riphah International Hospital, Islamabad, ICT, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Li S, Li Y, Liang Q, Yang WJ, Zi R, Wu X, Du C, Jiang Y. Effects of tele-exercise rehabilitation intervention on women at high risk of osteoporotic fractures: study protocol for a randomised controlled trial. BMJ Open. 2022 Nov 7;12(11):e064328. doi: 10.1136/bmjopen-2022-064328. PMID 36344002
- [Result] Rezaei MK, Torkaman G, Bahrami F, Bayat N. The effect of six week virtual reality training on the improvement of functional balance in women with type-I osteoporosis: A preliminary study. Sport Sci Health. 2023;19(1):185-194. doi: 10.1007/s11332-022-01018-8. Epub 2022 Nov 15. PMID 36408530
- [Result] Wei F, Hu Z, He R, Wang Y. Effects of balance training on balance and fall efficacy in patients with Osteoporosis: A systematic review and meta-analysis with trial sequential analysis. J Rehabil Med. 2023 May 17;55:jrm00390. doi: 10.2340/jrm.v55.4529. PMID 37194565